CLINICAL TRIAL: NCT06294093
Title: Differences Between Long Distance Road Runners and Treadmill Runners in Achilles Tendon Structure, Muscle Strength, Proprioception and Balance Performance
Brief Title: Differences Between Long Distance Road Runners and Treadmill Runners in Achilles Tendon Structure
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Zinman College of Physical Education and Sports Sciences (Other)
Responsible Party: Principal Investigator, Gali Dar, Principal Investigator, University of Haifa
Other Study IDs: 026/24
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Achilles Tendon Injury
Keywords: Achilles tendon; running

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treadmill group: healthy subjects who run regularly at least twice a week for half an hour, over 80% of the training on treadmill.
- road group: healthy subjects who run regularly at least twice a week for half an hour, over 80% of the training on road.

SUMMARY:
this study will investigate the structure of the Achilles tendon and functional tests in road runners compared to treadmill runners.

DETAILED DESCRIPTION:
Healthy runners (road and treadmill runners) who run regularly at least twice a week for half an hour, over 80% of the training on the treadmill or road, will be recruited for the study.

All subjects will fill out a demographic questionnaire for personal details (age, sex, height, weight, past injuries, training). Each participant will undergo functional tests in random order: 1. Examination of the morphology of the Achilles tendon - will be examined by ultrasound tissue characterized (UTC) 2. Balance test - Y Balance Test 3. Proprioception test - AMEDA device 4. Muscle strength test - manual dynamometer for testing gastrocnemius muscle strength. 5. Gastrocnemius muscle endurance test - single leg heel raise test until fatigue.

A comparison will be made between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* run regularly at least twice a week for half an hour,
* over 80% of the training on a treadmill or road

Exclusion Criteria:

* pain or injury to Achilles tendon during the 6 months, preventing running for at least 3 days.
* past Achilles tendon surgeries,
* sprained ankle in the last six months,
* lower limb and back pain while running
* participants who report running with minimalist shoes.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy runners who run on a regular basis, without injuries or pain during the last 6 months
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
ultrasound tissue characterized | baseline
  percentage of type 1,2,3,4 fibers within the tendon
Balance test | baseline
  Y Balance Test - composite score: sum of 3 reach directions in centimeters divided by 3 times the limb length then multiplied by 100
Proprioception test | baseline
  AMEDA device - scores between 0 and 1, A higher score represents better proprioception ability.
muscle strength test | baseline
  hand held dynamometer dynamometer assessment of Gastrocnemius muscle
endurance test gastrocnemius muscle | baseline
  number of single leg heel raise test until fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Prof., Principal Investigator — University of Haifa
Locations (1):
- The Academic College at Wingate, Netanya, Israel

REFERENCES:
- [Result] Dar G, Waddington G, Stern M, Dotan N, Steinberg N. Differences Between Long Distance Road Runners and Trail Runners in Achilles Tendon Structure and Jumping and Balance Performance. PM R. 2020 Aug;12(8):794-804. doi: 10.1002/pmrj.12296. Epub 2020 Jan 18. PMID 31762215